CLINICAL TRIAL: NCT00001580
Title: Tissue Acquisition for Molecular Diagnostics
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970138; 97-C-0138
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-03

CONDITIONS: Neoplasm
Keywords: Molecular Diagnostics; Ovary; Tissue Acquisition; cDNA Library; CGAP
MeSH Terms: conditions — Neoplasms

SUMMARY:
Acquisition of fresh tumor and normal tissue samples are necessary for the preparation of cDNA libraries, microarray chips, and tissue specific probes, and proteomics development and validation. This protocol will allow acquisition of samples at the time of tissue sampling for surgery, diagnostic tests, or therapeutic phereses. These samples will be forwarded without patient identifiers, pathology reports, or other labels. Tissue pathology will be verified within the Laboratory of Pathology and samples used strictly for CGAP and Proteomic Initiative indications.

DETAILED DESCRIPTION:
Acquisition of fresh tumor and normal tissue samples is necessary for the preparation of cDNA libraries, microarray chips, tissue specific probes, and proteomics development and validation. This protocol will allow acquisition of patient samples at the time of tissue sampling for surgery, diagnostic tests, or therapeutic phereses. These samples will be forwarded without patient identifiers, pathology reports, or other labels. Tissue pathology will be verified within the Laboratory of Pathology and samples used strictly for CGAP and Proteomic Initiative indications.

ELIGIBILITY:
INCLUSION CRITERIA:

All patients willing to sign the informed consent for whom tissue, blood or body fluids will be available are eligible.

Histopathologic diagnosis will be confirmed in the Laboratory of Pathology, National Cancer Institute and is not a criteria for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1997-06; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Emmert-Buck MR, Bonner RF, Smith PD, Chuaqui RF, Zhuang Z, Goldstein SR, Weiss RA, Liotta LA. Laser capture microdissection. Science. 1996 Nov 8;274(5289):998-1001. doi: 10.1126/science.274.5289.998. PMID 8875945
- [Background] Krizman DB, Chuaqui RF, Meltzer PS, Trent JM, Duray PH, Linehan WM, Liotta LA, Emmert-Buck MR. Construction of a representative cDNA library from prostatic intraepithelial neoplasia. Cancer Res. 1996 Dec 1;56(23):5380-3. PMID 8968089
- [Background] Emmert-Buck MR, Vocke CD, Pozzatti RO, Duray PH, Jennings SB, Florence CD, Zhuang Z, Bostwick DG, Liotta LA, Linehan WM. Allelic loss on chromosome 8p12-21 in microdissected prostatic intraepithelial neoplasia. Cancer Res. 1995 Jul 15;55(14):2959-62. PMID 7606709